CLINICAL TRIAL: NCT00629681
Title: Efficacy and Safety of Pregabalin in an Open-label, Non-comparative, Flexible-dose Trial With Diabetic Peripheral Neuropathy or Postherpetic Neuralgia
Brief Title: A Study of the Efficacy and Safety of Pregabalin for the Treatment of Diabetic Peripheral Neuropathy or Postherpetic Neuralgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081031
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2011-04

CONDITIONS: Painful Diabetic Neuropathy and Post Herpetic Neuralgia
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia, Postherpetic | interventions — Pregabalin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin capsules; initial dose of 75 mg twice daily for 4 days. Dose could be increased based on individual patient's response and tolerability to 150 mg twice daily from Day 4 onwards, with a further increase to 300 mg twice daily from Day 14 onwards if needed. Total duration of treatment was 28 days.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pregabalin for the treatment of diabetic peripheral neuropathy (DPN) or postherpetic neuralgia (PHN)

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of DPN or PHN
* Score on the Numeric Rating Scale of at least 4/10

Exclusion Criteria:

* Hospitalized patients
* Neurologic disorders unrelated to DPN or PHN or any severe pain that may confound the assessment of DPN- or PHN-related pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2004-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Correlation between global status (as measured by the Clinical Global Impression of Change [CGIC] and the Patient Global Impression of Change [PGIC]) and changes in pain, anxiety, and sleep parameters | Baseline to Week 4

SECONDARY OUTCOMES:
Mean sleep score from patient's daily sleep interference diary | 14 and 7 days before baseline, baseline, and Days 4, 7, 14, and 28
Change from baseline in mean sleep score from patient's daily sleep interference diary | End of treatment
Mean anxiety score from patient's daily anxiety diary | 14 and 7 days before baseline, baseline, and Days 4, 7, 14, and 28
Adverse events | 14 and 7 days before baseline, baseline, and Days 4, 7, 14, and 28
Change from baseline in Pain Treatment Satisfaction Scale (PTSS) 9 items score | End of treatment
Median time to pain response profile | Over the first week
CGIC and PGIC | End of treatment
Change from baseline in EuroQOL (as measures by EQ-5D) | End of treatment
Change from baseline in mean anxiety score from patient's daily anxiety diary | End of treatment
Change from baseline in Medical Outcomes Study (MOS)-Sleep Scale score | End of treatment
Course of mean pain score of patient's daily pain diary (NRS) | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- Germany (40):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Albstadt
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bielefeld
  - Pfizer Investigational Site, Celle
  - Pfizer Investigational Site, Deggingen
  - Pfizer Investigational Site, Duisburg
  - Pfizer Investigational Site, Erbach im Odenwald
  - Pfizer Investigational Site, Erfurt
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Gera
  - Pfizer Investigational Site, Göppingen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hemsbach
  - Pfizer Investigational Site, Hildesheim
  - Pfizer Investigational Site, Holle
  - Pfizer Investigational Site, Itzehoe
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Katzhütte
  - Pfizer Investigational Site, Leer
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Limburgerhof
  - Pfizer Investigational Site, Ludwigshafen
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, Lünen
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Marl
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Osnabrück
  - Pfizer Investigational Site, Recklinghausen
  - Pfizer Investigational Site, Senftenberg
  - Pfizer Investigational Site, Sinsheim
  - Pfizer Investigational Site, Surwold
  - Pfizer Investigational Site, Unterhaching
  - Pfizer Investigational Site, Veitsbronn
  - Pfizer Investigational Site, Weimar
  - Pfizer Investigational Site, Wiesbaden
  - Pfizer Investigational Site, Witten
  - Pfizer Investigational Site, Zwönitz

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081031&StudyName=A%20study%20of%20the%20efficacy%20and%20safety%20of%20pregabalin%20for%20the%20treatment%20of%20diabetic%20peripheral%20neuropathy%20or%20postherpetic%20neuralgia